CLINICAL TRIAL: NCT03644927
Title: Neurobiological Mediators of Self-Regulatory and Reward-Based Motivational Predictors of Exercise Maintenance in Chronic Pain and PTSD
Brief Title: Exercise Maintenance in Chronic Pain and PTSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended in 2020 due to Covid-19 policies, the study has now been terminated given recruitment and intervention challenges with the pandemic surge and end of funding.
Sponsor: Boston University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-37824; 1R21AT010293-01 (NIH)
Record Dates: First submitted 2018-08-17; First posted 2018-08-23 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-12

CONDITIONS: Chronic Low Back Pain; Posttraumatic Stress Disorder
Keywords: Veterans; Cardiopulmonary exercise testing; Exercise maintenance; Neuropeptide Y (NPY); Exercise-related intrinsic motivation; Exercise Self efficacy; Transtheoretical Model (TTM); Self-Determination Theory (SDT)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive exercise program (Experimental): Based on the "Active Physical Treatment Model" individuals with chronic pain are typically and primarily sedentary or physically deconditioned and need a progressive approach to work up to standard exercise prescriptions as defined by the American College of Sports Medicine. Thus, progressive exercise training can help to minimize the risk or occurrence of a range of exercise-related adverse medical events, particularly with the complex study population which will be starting at a sedentary level and therefore, may not be able to initially achieve the heart rate goals prescribed in standard exercise training protocols. The exercise prescription will be individually designed and geared toward an intensity manageable by the individual.
  Interventions: Behavioral: Progressive exercise training
- Waitlist Control (Active Comparator): The waitlist control participants will be fully screened for eligibility and asked to wait 12 weeks before beginning the 12-week progressive exercise program. They will be assessed again at the end of the 12-week waiting period. These patients will then be compared to patients in the experimental arm and then compared against their own waitlist control data after completing the 12-week exercise program. The exercise program that the waitlist control patients will participate in is identical to the experimental arm.
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: Progressive exercise training — The 12 week progressive exercise program gradually increases the walking/running intensity and length of exercise every 2 weeks for the first 6 weeks and then maintains the higher intensity level for weeks 7-12,. The exercise intensity is based on percentile targets defined by the baseline cardiopulmonary test (CPX test). Participants will be called at weeks 4 and 10 to assess and foster exercise motivation, using basic principles of motivational interviewing..
  Arms: Progressive exercise program
Behavioral: Waitlist Control — Participants will be screened for eligibility and if randomized into the waitlist control group. Wait list participants will wait for 12-weeks before they can participate in the progressive exercise training program. The 12 week progressive exercise program is identical to the one used in the intervention group. Specifically, the 12 week progressive exercise program gradually increases the walking/running intensity and length of exercise every 2 weeks for the first 6 weeks and then maintains the higher intensity level for weeks 7-12. The exercise intensity is based on percentile targets defined by the baseline cardiopulmonary test (CPX test). Participants will be called at weeks 4 and 10 to assess and foster exercise motivation, using basic principles of motivational interviewing.
  Arms: Waitlist Control

SUMMARY:
The primary purpose of the R21 is using an experimental medicine research approach to study whether a chronic, progressive-based exercise program will help Veterans suffering from chronic low back pain (cLBP) and PTSD achieve exercise maintenance, and shared symptom reduction, through neuropeptide Y mediated improvements in putative factors (self-regulation and reward sensitivity) known to improve exercise related self-efficacy and motivation.

DETAILED DESCRIPTION:
This study will compare the effects of a 3-month, individually prescribed progressive exercise training program on: 1) chronic low back pain (cLBP), depression and PTSD symptoms, and 2) neurobiological and related neuropsychological mechanisms by which our exercise-training paradigm may foster exercise maintenance. More specifically, the investigators hypothesize relationships between exercise-training associated augmentation of neuropeptide Y (NPY) system function and improved capacities for reward and self-regulation-neuropsychological capacities posited to underlie intrinsic motivation and self-efficacy, which in turn have been shown to predict exercise maintenance. This study will focus on Veterans with cLBP/PTSD. The study design includes a baseline, acute, cardiopulmonary exercise assessment (CPX) that will inform the exercise prescription for the 12-week "progressive exercise" training program, comprised of three 30-45 minute in clinic exercise sessions per week (walking or running--depending on the ability/capacity of the participant). All exercise sessions will be supervised by an exercise physiologist in the Clinical Studies Unit (CSU) at VA Boston Healthcare System. Intermittent telephone calls by the researchers will provide additional motivational support and problem solving. Implementation of the prescribed exercise regimen will also be supported by the use of heart rate and actigraph monitors programmed for the participant to achieve their prescribed heart rate range (HRR). Also, a "midpoint" and "endpoint" CPX assessment will track changes in NPY system function and delineate their impact on pain, depression and PTSD symptoms, as well as the factors proposed to foster exercise maintenance. All three CPX tests will be performed in accordance with guidelines published by the American College of Cardiology. Among Veterans with cLBP/PTSD, the investigators hypothesize that the capacity to release NPY in response to vigorous exercise (i.e., acute CPX testing) will be associated with improvements in pain, depression and PTSD symptoms, as well as the putative factors that predict exercise maintenance. Data from this R21 will be used to demonstrate feasibility and inform the further development of individually prescribed, motivationally based exercise regimens that could be used as adjuncts to cognitive and other therapeutic PTSD, depression or chronic pain interventions to reduce cLBP, depression and PTSD, as well as the negative consequences of these disorders over the long-term.

*Note: mandatory covid precautions due to the pandemic led to an initial suspension of all study activities in 2020 after just one of the consented enrolled participants was randomized into the 'progressive exercise' study arm. That participant completed only half of the 12 week intervention. In addition, this participant had one adverse event after a stress test which was determined to be unrelated to the study intervention. Despite intentions to resume the research, a decision was made to terminate the study in early 2022 given the recruitment and intervention challenges with the pandemic surge and the end of funding. No data wee collected related to any of the study outcome measures so no outcome measures are reported.

ELIGIBILITY:
Inclusion Criteria:

1. ICD-9 or ICD-10 diagnosis of chronic low back pain, as confirmed by the rehabilitation medicine doctor consulting to the study, and a confirmed comorbid psychiatric diagnosis of PTSD. More specifically, the CLBP/PTSD participant must meet for current chronic PTSD (>3 months) as assessed by the CAPS-5, 1-Month Diagnostic Version.
2. A medical history, physical examination, vital signs, EKG, and baseline laboratory studies, including urine toxicology screens and a negative urine pregnancy test (woman only), indicate that symptom-limited cardiopulmonary exercise stress (CPX) testing will be safe.
3. Women of child bearing capacity must agree to use effective contraception while participating; a urine pregnancy test performed on the morning prior to completing CPX testing will also be done.
4. Relatively sedentary at enrollment, as defined by the American College of Sports Medicine (i.e., performing less than 30 minutes/day and less than 150 minutes per week of moderate physical activity).
5. Free of medications and other substances (e.g., illicit drugs and alcohol) with effects that could hinder data interpretation for 2-6 weeks before the cold pressor test (CPT) and CPX testing depending on the medication and frequency of use (which must be cleared by the study Co-I and study MD, Dr. Rasmusson).
6. Psychotropic medications are allowed, as long as the participant has been stable on them for two months.
7. Tobacco product use is allowed; participants will not be required to lower or stop their dosage/intake; intensity of smoking will be monitored across the study via use of urine testing for cotinine (a long-lived metabolite of nicotine) at each test session. Regular morning nicotine users will be instructed to smoke/chew to satisfaction just prior to arriving at the Clinical Studies Unit for testing, which will be approximately 2-3 hours prior to performance of the CPT and CPX.
8. Using pain medications other than opiates provided none taken for 5 half-lives before CPT/CPX testing, generally about 24 hours.
9. Other anxiety or depressive disorders are permitted
10. May be involved in supportive psychotherapies as long as their participation has been stable for 3 months prior to study entry and remains stable throughout the course of the study
11. Can have a mild to moderate TBI, as determined by the BAT-L assessment.
12. Taking medications for chronic psychiatric or medical illnesses is allowed as long as the medications and medication dosing are stable for two months prior to participation in the study and remain stable throughout the 12 week exercise training protocol and final exercise test.

Exclusion Criteria:

1. A life threatening or acute physical illness (e.g., cancer), current schizophreniform illnesses, bipolar disorder, or active suicidal or homicidal ideation requiring clinical intervention.
2. Current or past alcohol and/or substance dependence (less than three months from date of screening assessment)
3. Current opiate pain medication use
4. Women who are or are planning to become pregnant within the next six months
5. Individuals seeking pain treatment such as surgical interventions or who have a neuropathic origin to their pain
6. Cannot tolerate exercising on a treadmill or on an upright bike due to chronic pain
7. A clinical history of coronary artery disease or positive stress test, uncontrolled cardiac arrhythmia, moderate-to-severe aortic stenosis, severe arterial hypertension (systolic >200 mmHg, diastolic>110 mm Hg) and more than first degree atrioventricular block
8. Severe TBI, as evidenced on the VA TBI screen and the BAT-L assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica R Scioli, PhD, Principal Investigator — Boston University
Locations (1):
- VA Boston Healthcare System, Jamaica Plain, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scioli ER, Smith BN, Whitworth JW, Spiro A, Esterman M, Dutra S, Bogdan KM, Eld A, Rasmusson AM. Moderated mediation for exercise maintenance in pain and posttraumatic stress disorder: A randomized trial. Health Psychol. 2020 Sep;39(9):826-840. doi: 10.1037/hea0000876. PMID 32833484

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 92 potential participants were identified. 37.4% (n=34/92) were determined to be ineligible, 7.7% were loss to follow-up prior to signing consent, 3.2% had unknown status, 34.7% were in the process of being scheduled for their screening, 20.9% (n=19) had a screening visit scheduled and 11 of those were screened and provided signed consent.
Pre-assignment Details: Only one of the 11 consented participants was randomized into a study arm, the other 10 were not randomized prior to study termination. The 'progressive exercise' arm participant only completed 6 of the 12 weeks intervention before the study was terminated nut did not provide any outcome measure data and due to concerns over confidentiality no baseline data for that one participant will be reported.
Groups:
- Progressive Exercise Program: The 12 week progressive exercise program gradually increases the walking/running intensity and length of exercise every 2 weeks for the first 6 weeks and then maintains the higher intensity level for weeks 7-12. The exercise intensity is based on percentile targets defined by the baseline cardiopulmonary test (CPX test). Participants will be called at weeks 4 and 10 to assess and foster exercise motivation, using basic principles of motivational interviewing.
- Waitlist Control: Wait list participants will wait for 12 weeks before they can participate in the progressive exercise training program. The 12-week progressive exercise program is identical to the one used in the intervention group. Specifically, the 12-week progressive exercise program gradually increases the walking/running intensity and length of exercise every 2 weeks for the first 6 weeks and then maintains the higher intensity level for weeks 7-12.
Period: Overall Study
Arm/Group | Progressive Exercise Program | Waitlist Control
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — The single subject in this arm didn't complete the 12 weeks intervention before study termination. | 1 | 0

BASELINE CHARACTERISTICS:
Population: Since only one participant was randomized into a study arm. The baseline characteristics are provided for all 11 consented participants aggregated into a single group to protect confidentiality of the single randomized particiapnt.
Groups:
- All Participants: All enrolled participants are aggregated into one group since only one participant was randomized into one of the 2 study arms prior to termination of the study.
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 48.8 [29 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3
  Caucasian | 6
  Asian | 1
  Hispaic | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Transtheoretical Model of Exercise: Stages of Change (Short-form)
Description: This 4-item continuous measure categorizes stages of behavioral change based on the Transtheoretical Model (TTM) stages (precontemplation, contemplation, preparation, action and maintenance), specifically in the context of exercise behavior change. Each stage reflects a different level of readiness to exercise, where precontemplation means that the patient is not actively considering exercise behaviors, whereas a patient in the maintenance stage has been actively exercise regularly (3 times per week for 50 minutes minimum) for at least the past 6 months. Scoring for this measure is determined by YES or NO answers provided to questions about exercise behaviors that patients are currently doing or intend to do in the near future. For example, if patients answer YES to the first question "Do you currently engage in regular exercise (at least 3 times per week for 50 or more minutes per session)?", then the patient could either be in the action or maintenance stage of exercise.
Time Frame: Eligibility/screening, baseline, 6 week, and 12 week
Population: Only one of the 11 consented participants was randomized into a study arm, the other 10 were not randomized prior to study termination. The 'progressive exercise' arm participant only completed 6 of the 12 weeks intervention before the study was terminated nut did not provide any outcome measure data and due to concerns over confidentiality no baseline data for that one participant will be reported.
Groups:
- Progressive Exercise Program: The 12-week progressive exercise program gradually increases the walking/running intensity and length of exercise every 2 weeks for the first 6 weeks and then maintains the higher intensity level for weeks 7-12. The exercise intensity is based on percentile targets defined by the baseline cardiopulmonary test (CPX test). Participants will be called at weeks 4 and 10 to assess and foster exercise motivation, using basic principles of motivational interviewing.
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: ActiGraph Monitor
Description: Objective verification of exercise compliance over time
Time Frame: over the course of 12 weeks of exercise training
Population: as for outcome 1
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: West Haven Yale Multidimensional Pain Inventory - Pain Interference
Description: The West Haven Yale Multidimensional Pain Inventory (WHYMPI) has been demonstrated to be applicable across a variety of clinical pain conditions, and this subscale focuses on pain interference. Participants identify a "significant other" defined as a person with whom the participant feels closest to by checking off one of 7 descriptive terms that best represents the relationship with this person and if the participant shares a living space with that person. Next are 20 items about the impact of pain on the participant's life and are scored on a 7-point scale from 0 to 6. Some questions are reverse coded and a higher overall score indicates greater pain interference. Some anchors for 0 to 6 include "No pain/Very intense pain," "No interference/Extreme interference," "No change/Extreme change," "Not at all supportive/Extremely supportive," and "Extremely low mood/Extremely high mood."
Time Frame: Eligibility/Screening, baseline, 6 week, 12 week
Population: as for outcome 1
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Clinician-Administered PTSD Scale-5
Description: The CAPS is the gold standard in PTSD assessment. The CAPS-5 is a 30-item structured interview that can be used to make a current (past month) diagnosis of PTSD, lifetime diagnosis of PTD, and assesses PTSD symptoms over the past week. The patient identifies a Criterion A index trauma and the assessor combines information about frequency and intensity of each item into a single severity rating. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: Criterion B (items 1-5); Criterion C (items 6-7); Criterion D (items 8-14); and, Criterion E (items 15-20). A symptom cluster score may also be calculated for dissociation by summing items 19 and 20. Criterion items are scored 0 to 4 (Absent to Extreme/incapacitating) and summed up. Higher scores indicate greater severity of PTSD.
Time Frame: Eligibility/screening and 12 week
Population: as for outcome 1
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Self-Efficacy for Exercise
Description: This 6-item scale is used to determine confidence in one's ability to exercise. Total score is calculated by summing the responses to each question. Participants rate self-efficacy to exercise in specific situations on 5-point scale from Not at all Confident to Completely Confident. A higher score indicates higher self-efficacy for exercise.
Time Frame: Eligibility/Screening, baseline, 6 week, 12 week
Population: as for outcome 1
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Generalized Self-Efficacy Scale
Description: This revised10-item scale taps into a global sense of self-efficacy, or belief by an individual in his or her ability (e.g., "I can always solve difficult problems if I try hard enough, " and "I can usually handle whatever comes 66-68 This 10-item self-report scale assesses habitual use of two common strategies to alter emotion captured on two sub-scales: cognitive reappraisal and expressive suppression. Items are rated on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree).
Time Frame: Eligibility/Screening, baseline, 6 week, 12 week
Population: as for outcome 1
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Temporal Experience of Pleasure Scale
Description: This 18-item self-report measure uses a Likert-like scale (1-6) to assess reward sensitivity to specific experiences that are either anticipatory (the night before a major holiday) or consummatory (chocolate chip cookie). Participants rate from 1 (very false for me) to 6 (very true for me) when presented statements about how one might react to specific rewarding stimuli. Scores are added together and greater score represent higher anticipation of a reward, higher enjoyment when presented a tangible reward, a greater total score (subscales added) represents a higher sensitivity to rewarding stimuli.
Time Frame: Eligibility/Screening, baseline, 6 week, 12 week
Population: as for outcome 1
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Effort Expenditure for Rewards Task
Description: This computerized (Matlab) task (for which scripts have been obtained from the developer for study use) captures willingness to expend effort for rewards. EEfRT scores have been inversely related to anhedonia. The task has been validated in healthy college students and adults with major depression and schizophrenia.
Time Frame: Eligibility/Screening, baseline, 6 week, 12 week
Population: as for outcome 1
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Neuropeptide-Y
Description: The blood plasma will be collected in EDTA tubes and placed immediately on wet ice; it will be spun within 20 minutes of collection at 3000 rpm for 15 minutes in a refrigerated centrifuge before aliquoting into tubes for storage at -70 degrees C until assays of the neurosteroids/peptides of interest are performed. Plasma NPY will be measured by radioimmunoassay (RIA) as previously described (Rasmusson et al., 2000).
Time Frame: Baseline, 6 week, 12 week
Population: as for outcome 1
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Go/No-Go Task
Description: This computerized task measures response inhibition. Participants are asked to respond to certain ("go") stimuli and make no response "no-go" stimuli, while maintaining speed and accuracy The main dependent measure is the commission error rate making a "go" response to "no-go" trials.
Time Frame: Baseline, 6 week, 12 week
Population: as for outcome 1
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Exercise Motivation Scale
Description: This 31-item scale is used to determine extrinsic and intrinsic variants of exercise motivation based on Self-Determination Theory. Participants rate statements about personal motivation from 1 (strongly disagree) to 6 (strongly agree), depending on how strongly the participant relates to each item. Higher scores on specific items reflect the major sources of the participant's motivation to exercise. For example, higher scores on items 2, 10, 15, and 27 indicates intrinsic motivation to learn more about/from exercising.
Time Frame: Eligibility/Screening, baseline, 6 week, 12 week
Population: The study was terminated prior to randomization into the study arms and no participant received any intervention.
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Beck Depression Inventory
Description: The Beck Depression Inventory-II (BDI-II) is a well-validated 21-item self-report measure of depressive symptom severity. It yields a total score and subscale scores for depressive cognitive and somatic symptoms. BDI-II items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is calculated by adding the sums of both subscales, with 0-13 indicating minimal depression, 14-19 indicating mild depression, 20-28 indicating moderate depression, and 29-63 indicating severe depression.
Time Frame: Eligibility/Screening, baseline, 6 week, 12 week
Population: as for outcome 1
Arm/Group | Progressive Exercise Program | Waitlist Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the 6 weeks that one participant received the study intervention prior to study termination. In addition prior to randomization two participants had an adverse event during the rigorous and conservative screening process and they were not allowed to proceed to the intervention. One participant felt nauseous and had a headache and the other had abnormal EKG findings and a positive history for cardiac issues.
Groups:
- Progressive Exercise Program: Only one participant was randomized into this study arm prior to study termination and they only completed half [6 out of the 12 week] of the study intervention prior to study termination.
Arm/Group | Progressive Exercise Program
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progressive Exercise Program (N=11)
Nausea (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Cardiac abnormalities (Cardiac disorders) | 1 (1) — During Screening an abnormal EKG was obtained and a history of previous cardiac issues reported by participant.

LIMITATIONS AND CAVEATS:
Only one of the 11 consented participants was randomized into a study arm, the other 10 were not randomized prior to study termination. The 'progressive exercise' arm participant only completed 6 of the 12 weeks intervention before the study was terminated so no data were collected for any of the outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT03644927/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT03644927/ICF_001.pdf